CLINICAL TRIAL: NCT02164188
Title: The Flourishing Project: Evaluation of the Effectiveness of a Well-being Program in the Personal and Relational Dimensions
Brief Title: The Flourishing Project: Evaluation of the Effectiveness of a Well-being Program
Acronym: Flourishing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Elisa Kozasa, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIAE_Florescer
Record Dates: First submitted 2014-04-29; First posted 2014-06-16 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Emotional Stress
Keywords: Stress; Well-being; Functional magnetic resonance imaging; Positive psychology
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Initially this control group will not receive an intervention (wait list). After 8 weeks this goup will receive the Flourishing protocol (cross over).
- Flourishing protocol (Experimental): This group will receive the intervention Flourishing protocol and after that it will not receive any other intervention (cross over).
  Interventions: Behavioral: Flourishing protocol

INTERVENTIONS:
Behavioral: Flourishing protocol — This intervention is based on relaxation, well-being promotion, meditation practices, positive psychology principles. The format is 1hour and half meetings during 8 weeks, and daily practices. MP3 audios are presented for daily practices.
  Arms: Flourishing protocol

SUMMARY:
This protocol proposes a well-being program based on meditation and Positive Psychology principles such as human development, the improvement of virtues, quality of life and well-being. The investigators hypothesize that this program may promote well-being and reduce stress related problems in the participants. Objectives: To evaluate the efficacy of a well-being program in a sample of managers who work in a company (Natura Inovação/Cosméticos ) and health care professionals who work in a hospital (Hospital Israelita Albert Einstein) as well as its implication in the work environment. Methods: Sixty managers from Natura Inovação/Cosméticos and 60 health professionals from Hospital Israelita Albert Einstein will be recruited. The participants will be randomized in two groups of 30 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI).

DETAILED DESCRIPTION:
Introduction: Stress related disorders may lead to mental disorders as well as cardiovascular problems. They may also result in absenteeism and less productivity in companies. This protocol proposes a well-being program based on meditation and Positive Psychology principles such as human development, the improvement of virtues, quality of life and well-being. The investigators hypothesize that this program may promote well-being and reduce stress related problems in the participants. Objectives: To evaluate the efficacy of a well-being and quality of life program in a sample of managers who work in a company (Natura Inovação/Cosméticos ) and health care professionals who work in a hospital (Hospital Israelita Albert Einstein) as well as its implication in the work environment. Methods:Sixty participants from Natura Inovação/Cosméticos and 60 health professionals from Hospital Israelita Albert Einstein will be recruited. The participants will be randomized in two groups of 30 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI). This is a cross-over study. After the first evaluation GI will participate in the Flourishing Program for 8 weeks and the GC will be a wait-list group in this period of time. After that, there is a second evaluation of the participants and the GC will receive the intervention (Flourishing Program). GI will not receive any intervention during this new period of 8 weeks. A final evaluation will happen after that. The participants will fill in questionnaires (to evaluate depression, anxiety, stress, positive and negative affects, sleep quality, self-compassion, mindfulness, virtues, values, happiness, psychological well-being) and will be clinically examined; their blood sample will be collected (for the dosage of health related biomarkers) and also saliva for cortisol measures. They will perform structural and functional neuroimaging exams (emotional and cognitive paradigms) and their physiological measures such as skin conductance will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female aging from 25 to 60
* Managers from Natura Company or healthcare professionals from Hospital Israelita Albert Einstein

Exclusion Criteria:

* Sever mental or physical diseases
* For fMRI we will exclude participants who don´t match the criteria to undergoing this exam.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04-03 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress | (baseline, 3 months, 6 months)
  Lipp Stress Inventory; Perceived Stress Scale
Changes in well-being | baseline, 3 months, 6 months
  WHOQOL-bref (World Health Organization Quality of Life Questionnaire with 26 questions); Well-being at work scale; Psychological well-being scale.

SECONDARY OUTCOMES:
Change in cortisol levels | Baseline; 3 months; after 6 months
  Saliva will be collected to measure cortisol levels: 7-9 am, 4-5 pm, 11-12 pm.

OTHER OUTCOMES:
Changes in brain function | Baseline; 3 months; 6 months
  Functional magnetic resonance imaging exams: emotional (International Affective Pictures System) and cognitive paradigms (Stroop Word Color Task and N-back).
Changes in anxiety symptoms | baseline, 3 months,6 months
  Beck Anxiety Inventory
Changes in depression symptoms | baseline, 3 months, 6 months
  Beck Depression Inventory
Changes in mindfulness | baseline, 3 months, 6 months
  Mindful Awareness Attention Scale
Changes in Positive and Negative Affect | baseline, 3 months, 6 months
  PANAS questionnaire
Changes in Psychological capital | baseline, 3 months, 6 months
  Psychological Capital Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Kozasa, PhD, Principal Investigator — Instituto do Cérebro- Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- See also: A yoga and compassion meditation program reduces stress in familial caregivers of Alzheimer's disease patients. — http://www.ncbi.nlm.nih.gov/pubmed/23690846
- See also: Meditation training increases brain efficiency in an attention task. — http://www.ncbi.nlm.nih.gov/pubmed/21763432